CLINICAL TRIAL: NCT05949658
Title: Safer mTOR Inhibition for Human Geroprotection
Brief Title: Rapalog Pharmacology (RAP PAC) Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-0275; 1U01AG081482-01 (NIH); SMPH/MEDICINE/GER-AD DEV (Other: UW Madison); Protocol Version 1/30/2025 (Other: UW Madison)
Record Dates: First submitted 2023-06-26; First posted 2023-07-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Aging
Keywords: Rapamycin; Rapamycin analog; mTOR; mTOR inhibitor; sirolimus; everolimus; rapamune
MeSH Terms: interventions — Sirolimus; Everolimus

STUDY DESIGN:
Intervention Model Description: The Bayesian Optimal Interval Design (BOIN) will be used to perform a phase I, dose finding trial in healthy older men and women (55-89yrs) for the mTOR inhibitors sirolimus and everolimus. Middle-aged to older adults will be treated with either sirolimus or everolimus for 6 weeks. All participants will take one capsule weekly. This dose escalation trial will begin with two cohorts, each consisting of 3 male and 3 female participants. The first two cohorts will take a weekly 5mg dose of sirolimus or a weekly 5mg dose of everolimus. Researchers will enroll for both arms of the study concurrently. Participants will be informed that they will be allocated to the next available opening that works with their schedule, which could be either everolimus or rapamycin. The dose can be escalated/de-escalated from the current dose based on the rate of dose limited toxicity (DLT) at the end of the 6-week intervention for each cohort. The 15mg dose will be the highest dose possible in this trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sirolimus (Experimental): 1mg tablets of sirolimus that total the assigned dose
  Interventions: Drug: Sirolimus
- Everolimus (Experimental): 1mg tablets of everolimus that total the assigned dose
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Sirolimus — 5mg, 10mg, or 15mg once weekly sirolimus
  Other Names: Rapamycin
  Arms: Sirolimus
Drug: Everolimus — 5mg, 10mg, or 15mg once weekly everolimus
  Arms: Everolimus

SUMMARY:
The objective of RAP PAC is to identify safe and effective weekly dose(s) for the mTOR inhibitors sirolimus and everolimus that intervene on the underlying fundamental biology of aging. Participants who are 55-89 years old that are free of overt chronic diseases will be assigned to either 6 weeks of sirolimus or everolimus (5 mg, 10 mg, or 15 mg once per week). The investigators will complete the everolimus arm first and then subsequently complete the sirolimus arm of the study. Total time on study would be up to 17 weeks to complete baseline and follow up visits.

DETAILED DESCRIPTION:
The mTOR inhibitor rapamycin and rapamycin analogs (rapalogs) extend healthspan and/or lifespan in multiple model systems. However, the risk of adverse events and dose limiting toxicities in humans have thus far precluded the long-term prophylactic use of mTOR inhibitors as a therapy for aging and age-related diseases. The pharmacokinetics and pharmacodynamics (PK/PD) data for mTOR inhibitors in older adults is currently unknown and has prevented the identification of a safe dosage that could maximize health-span extension and minimize adverse effects.

RAP PAC will identify a recommended phase 2 trial dose for sirolimus and everolimus in older men and women by performing a phase 1, dose finding study that evaluates PK/PD, safety and tolerability, and mTOR signaling using conventional as well as novel approaches. Overall, the investigators will pair comprehensive molecular and pharmacologic approaches to evaluate PK/PD in humans and identify dosing regimens that safely inhibit mTOR complex 1 (mTORC1) to intervene in the biology of aging.

ELIGIBILITY:
Inclusion Criteria:

* Middle-age adults free of overt chronic disease
* Willing to provide informed consent
* Willing to comply with all study procedures and be available for the duration of the study
* Able to use and be contacted by telephone
* Ability to take oral medication
* Not planning to change diet or physical activity status
* Adequate organ function as indicated by standard laboratory tests: hematology (complete blood count), and clinical chemistry
* Males must agree to avoid impregnation of women during and for four weeks after completing study visits through use of an acceptable method of contraception

Exclusion Criteria:

* Heart disease (history, abnormal ECG)
* Cerebrovascular disease (history)
* Cancer or less than 5 years in remission (history)
* Chronic respiratory disease (history, FEV1/FVC < 70, FEV1 < 80% predicted)
* Chronic liver disease (history, abnormal blood liver panel, ALT >104 IU/L, AST >80 IU/L)
* Diabetes (history, HbA1C ≥ 6.5, fasting blood glucose≥126 mg/dl, OGTT ≥ 200 mg/dl at 2 hrs.)
* Alzheimer's (history)
* Chronic kidney disease (history, abnormal blood kidney panel including serum creatinine>1.4, eGFR≤60 ml/min/1.73m2)
* Problems with bleeding, on medication that prolongs bleeding time (if subject cannot safely stop prior to biopsy)
* Taking azathioprine (Imuran), cyclosporine (Gengraf, Neoral, Sandimmune), dexamethasone (Decadron, Dexpak), methotrexate (Rheumatrex, Trexall), prednisolone (Orapred, Pediapred, Prelone), prednisone (Sterapred), sirolimus (Rapamune), and tacrolimus (Prograf) or other medications proposed to lower the immune system
* Taking strong or moderate CYP3A4 and/or P-glycoprotein (PgP) inhibitors such as ketoconazole, itraconazole, clarithromycin, atazanavir, nefazodone, saquinavir, telithromycin, ritonavir, indinavir, nelfinavir, voriconazole, amprenavir, fosamprenavir, aprepitant, erythromycin, fluconazole, verapamil, diltiazem
* Taking strong CYP3A4 activators such as phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital
* Subjects who are not willing to restrict the use of grapefruit, grapefruit juice, cannabidiol (CBD) and other foods/substances that are known to inhibit cytochrome P450 and PgP activity and may increase everolimus exposures and should be avoided during treatment
* Subjects who are not willing to restrict the use of St. John's Wort (Hypericum perforatum) because it may decrease everolimus exposure unpredictably.
* Subjects who are not willing to avoid blood donations 8 weeks prior to the first visit and 8 weeks after the last visit
* Low white-blood cell count (<4,000 cell/µL)
* History of stomatitis or ulcers in the mouth
* Those on glucose lowering drugs
* Participating in intensive exercise training program (high to moderate intensity exercise greater than 150 minutes per week) or planning to start new exercise program during study period
* Tobacco use
* Allergies to lidocaine, sirolimus, or everolimus
* Subjects currently enrolled in other clinical trials. Subjects may be eligible after a washout period that will be reviewed on a case-by-case basis.
* Individuals with limited English proficiency
* Subjects who are planning to have elective surgery 12 weeks prior to or during the intervention

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicities (DLTs) | Through study completion, an average 3 years
  A recommended phase 2 dose (RP2D) will be determined through evaluating dose limiting toxicities (DLT), which is defined as ≥Grade 2 adverse event following CTCAE v6.0.

SECONDARY OUTCOMES:
Time course of drug concentration in blood | First dose to 168 hours post dose
  Using PK parameters of Peak Plasma Concentration (Cmax, Cmin), determine duration of concentration of drug in blood measured pre dose, and 0.5, 1.5, 4, 48, and 168 hours post dose
Time course of drug concentration in blood | First dose to 168 hours post dose
  Using PK parameters of Area under the plasma concentration versus time curve (AUC, T1/2), determine duration of concentration of drug in blood measured pre dose, and 0.5, 1.5, 4, 48, and 168 hours post dose
Change in mTOR signaling in blood and muscle | 0 (pre-intervention) and 6 weeks (post-intervention)
  To be evaluated through immunoblotting and immunoprecipitation
Change in concentration of metabollites | 0 (pre-intervention) and 6 weeks (post-intervention)
  Metabolomics: Change in concentration of blood and/or skeletal muscle metabolites as assessed by liquid chromatography mass spectrometry
Change in concentration of lipid species | 0 (pre-intervention) and 6 weeks (post-intervention)
  Lipidomics: Change in the concentration of lipid species in blood and/or skeletal muscle as assessed by liquid chromatography mass spectrometry
Change in transcriptome | 0 (pre-intervention) and 6 weeks (post-intervention)
  Change in skeletal muscle and whole blood transcripts assessed via RNA sequencing
Change in glucose tolerance | 0 (pre-intervention) and 6 weeks (post-intervention)
  Assess change in glucose tolerance by area under the curve
Change in whole body insulin sensitivity | 0 (pre-intervention) and 6 weeks (post-intervention)
  Insulin sensitivity as assessed by the Matsuda Index.
Change in glucose variability | 0 (pre-intervention) and 6 weeks (post-intervention)
  Glucose Variability will be assessed via continuous glucose monitoring during two occasions during weeks 0, and 6 by measuring the change in range.
Change in glucose variability | 0 (pre-intervention) and 6 weeks (post-intervention)
  Glucose Variability will be assessed via continuous glucose monitoring during two occasions during weeks 0, and 6 by measuring the change in total standard deviation.
Change in glucose variability | 0 (pre-intervention) and 6 weeks (post-intervention)
  Glucose Variability will be assessed via continuous glucose monitoring during two occasions during weeks 0, and 6 by measuring the change in mean daily differences (MODD).
Change in glucose variability | 0 (pre-intervention) and 6 weeks (post-intervention)
  Glucose Variability will be assessed via continuous glucose monitoring during two occasions during weeks 0, and 6 by measuring the change in the overall net glycemic action over a 4-h and 8-h period (CONGA4; CONGA8).
Change in insulin resistance | 0 (pre-intervention) and 6 weeks (post-intervention)
  Measured by change in homeostatic model of insulin resistance (HOMA-IR).

CONTACTS AND LOCATIONS:
Overall Officials: Adam Konopka, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers years after the completion of the study endpoints by contacting Dr. Adam Konopka or the NIA BioBank Repository.